CLINICAL TRIAL: NCT04741945
Title: STOP-LEUKEMIA: Repurposing Metformin As a Leukemia-preventive Drug in CCUS and LR-MDS
Brief Title: Repurposing Metformin As a Leukemia-preventive Drug in CCUS and LR-MDS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kirsten Grønbæk (Other)
Collaborators: Steno Diabetes Center Copenhagen (Other); Zealand University Hospital (Other); Van Andel Research Institute (Other); Herlev Hospital (Other); Technical University of Denmark (Other); Region Hovedstadens Apotek (Other Government); University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Kirsten Grønbæk, Professor, MD, DMSc, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STOP-LEUKEMIA
Record Dates: First submitted 2021-01-19; First posted 2021-02-05 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Preleukemia; Myelodysplastic Neoplasm; Cytopenia; Preleukemic Anemia
Keywords: Metformin; Myelodysplastic Neoplasm; Clonal Cytopenia of Undetermined Significance; Safety; Feasibility; Bone Marrow Adipose Tissue; Gut Microbiota; Intestinal Permeability
MeSH Terms: conditions — Preleukemia; Anemia, Refractory, with Excess of Blasts; Cytopenia | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Metformin (Experimental): 2000 mg/day metformin for 12 months.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — 2000 mg/day metformin for 12 months (1000 mg b.i.d.) with a slow up-titration six weeks prior to full dose treatment.

SUMMARY:
This is a single-arm pilot study of the feasibility and safety of metformin in patients with clonal cytopenia of undetermined significance (CCUS) or lower-risk myelodysplastic neoplasms (LR-MDS).

DETAILED DESCRIPTION:
The research plan is divided into three work packages (WP):

WP0: Bone Marrow Adipose Tissue, Gut Microbiota, and Intestinal Permeability in CCUS and LR-MDS Patients.

The aim of WP0 is to investigate biological features which the investigators hypothesize to be of pathogenetic relevance for MDS progression and may be possible targets of metformin treatment. For this purpose, 20 elderly (≥60 years) healthy controls will be included for comparison to patients with CCUS or LR-MDS from WP1.

The primary objectives are to investigate 1) the abundance and properties of bone marrow adipose tissue (BMAT) and bone marrow (BM) adipocytes, and 2) the gut microbiota and intestinal permeability of patients with CCUS or LR-MDS compared to age-, sex- and body mass index (BMI)-matched healthy controls. Secondary objectives are to characterize DNA methylation and hydroxymethylation (5-mC and 5-hmC) patterns, and hormone and cytokine levels in BM plasma from healthy controls and patients with CCUS or LR-MDS.

WP1: Safety, feasibility, and mechanisms of action of metformin in patients with CCUS or LR-MDS.

In this WP up to 40 patients with CCUS or LR-MDS will receive metformin 2000 mg daily or their maximum tolerated dose (MTD) for 12 months. The aim of WP1 is to investigate safety of metformin and feasibility of the protocol in patients with CCUS or LR-MDS. Potential mechanisms of anti-leukemic action of metformin will also be explored in order to identify a suitable outcome measure and estimate standard deviation of the outcome measure. All in order to inform the design of a future phase 3 RCT of the efficacy of metformin in CCUS and LR-MDS patients. Endpoints of WP1 are specified in the corresponding section.

WP2: Safety and efficacy of metformin compared to placebo. The primary objective of WP2 is to compare safety and preliminary efficacy of metformin in patients with CCUS or LR-MDS to a cohort of patients with CCUS or LR-MDS receiving placebo in context of our EVI-2 randomized, controlled pilot study (NCT03999723).

Data and samples from approximately 50 historical controls will be included from the EVI-2 study in which participants were randomized to receive placebo or oral vitamin C supplement for 12 months.

ELIGIBILITY:
Patients are eligible to be included in WP1 if they meet all of the following criteria:

Inclusion criteria:

* A diagnosis of:

  * LR-MDS according to the revised international prognostic scoring system (IPSS-R), i.e., very low- or low-risk disease (IPSS-R score ≤3) in addition to a bone marrow blast percentage <5 OR
  * CCUS defined as the presence of somatic mutation(s) or cytogenetic abnormality not diagnostic of MDS or any other malignancy in the context of persistent cytopenia (>6 months) with other common causes of cytopenia ruled out in the setting of bone marrow morphology that is not diagnostic of MDS or any other malignancy, and hematolytic conditions have been ruled out. Peripheral blood cytopenia is defined as hemoglobin (hgb) <11.3 g/dL (7 mmol/L) in women and hgb <12.9 g/dL (8 mmol/L) in men, platelet count <150 x 109/L, or neutrophil count <1.8 x 109/L
* Menopause, if being a female, defined as females >45 years of age who have experienced amenorrhea for minimum 12 months, without any other obvious pathological or physiological cause
* ≥18 years of age
* Written informed consent
* Willingness to comply with mandatory aspects of the protocol
* Ability to swallow pills

Exclusion criteria:

* Any prior treatment with metformin
* A diagnosis of diabetes mellitus
* Therapeutic radiation, immunosuppressive therapy (with the exception of corticosteroids), or chemotherapy within the past year
* Treatment with granulocyte colony-stimulating factor within the past 30 days
* Prior therapy with hypomethylating agents (i.e., azacitidine, decitabine)
* eGFR <45 mL/min
* Performance status according to the Eastern Cooperative Oncology Group >2
* Other active malignancy within the past five years
* Uncontrolled comorbidity including impaired hepatic function (total serum bilirubin >1.5 × upper limit of the normal range (ULN), serum alanine transaminase >3 × ULN), chronic hepatitis with decompensated cirrhosis, disabling psychiatric disease, severe neurologic disease, uncontrolled metabolic disease, or severe cardiac disease (NYHA class 3-4)

An eGFR calculation performed up to one month prior to inclusion may be used to assess renal function. If such an assessment is not available, it is performed at screening.

Healthy volunteers are eligible to be included in WP0 if they meet all of the following criteria:

Inclusion criteria:

* Healthy individuals matched on age, sex, and BMI, if possible, to individual patient participants in WP1
* Written informed consent
* Willingness to comply with mandatory aspects of the protocol

Exclusion criteria:

* Use of metformin within the past 3 years
* A diagnosis of diabetes mellitus, rheumatological disorders, autoimmune diseases or other inflammatory disorders, celiac disease, inflammatory bowel disease, or other gastrointestinal disorders or symptoms
* Treatment with immunosuppressive drugs (with the exception of corticosteroids) or chemotherapy within the past year or antibiotics within the past 6 months
* Any contraindications to MRS

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by the number of serious adverse events including any suspected unexpected serious adverse reactions | From inclusion to 12 months of study treatment
  To assess safety of metformin treatment in this off-label indication by the type, grade, and number of adverse events and serious adverse events including any suspected unexpected serious adverse reactions in the patients.
Safety as assessed by median maximum tolerated dose in mg/day | From inclusion to 12 months of study treatment
  To assess safety of metformin treatment in this off-label indication by median maximum tolerated dose and a description of any changes in individual medication doses.
Feasibility as assessed by rates of recruitment/refusal rates | From inclusion to 12 months of study treatment
  To assess feasibility of the study protocol in terms of recruitment and refusal rates.
Feasibility as assessed by 12 months follow-up, i.e., study completion, rate | From inclusion to 12 months of study treatment
  To assess feasibility of the study protocol in terms of rate of study completion.
  To assess safety of metformin treatment in this off-label indication by the type, grade, and number of adverse events and serious adverse events including any suspected unexpected serious adverse reactions in the patients; drop-out rates; and a description of any changes in individual medication doses including median maximum tolerated dose.
Feasibility as assessed by rate of compliance to protocol procedures | From inclusion to 12 months of study treatment
  To assess feasibility of the study protocol in terms of rate of adherence to protocol procedures (study medication and study procedures).

SECONDARY OUTCOMES:
Interim efficacy: Mutational burden as assessed by change in variant allele frequency | From inclusion to 12 months of study treatment
  Change in variant allele frequency (ΔVAF) by next generation sequencing (NGS)
Interim efficacy: Patient-reported outcome measures based on the EORTC QLQ-C30 | From inclusion to 4 months of study treatment
  Change in patient-reported outcome measures (PROM), based on the validated European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30).
Interim efficacy: Patient-reported outcome measures based on the EORTC QLQ-C30 | From inclusion to 12 months of study treatment
  Change in patient-reported outcome measures (PROM), based on the validated European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30).
Interim efficacy: Patient-reported outcome measures based on the SF-36 | From inclusion to 4 months of study treatment
  Change in patient-reported outcome measures (PROM), based on the validated Short Form 36 Health Survey Questionnaire (SF-36).
Interim efficacy: Patient-reported outcome measures based on the SF-36 | From inclusion to 12 months of study treatment
  Change in patient-reported outcome measures (PROM), based on the validated Short Form 36 Health Survey Questionnaire (SF-36).
Interim efficacy: Patient-reported outcome measures based on the EQ-5D | From inclusion to 4 months of study treatment
  Change in patient-reported outcome measures (PROM), based on the validated European Quality of Life Five Dimension questionnaire (EQ-5D).
Interim efficacy: Patient-reported outcome measures based on the EQ-5D | From inclusion to 12 months of study treatment
  Change in patient-reported outcome measures (PROM), based on the validated European Quality of Life Five Dimension questionnaire (EQ-5D).
Interim efficacy: Bone marrow adipose tissue as assessed by MR spectroscopy ratio of adipose tissue and water phase | From inclusion to 4 months of study treatment
  Change in bone marrow adipose tissue (BMAT) content in bone marrow (BM) measured by MR spectroscopy
Interim efficacy: Bone marrow adipose tissue as assessed by MR spectroscopy ratio of adipose tissue and water phase | From inclusion to 12 months of study treatment
  Change in bone marrow adipose tissue (BMAT) content in bone marrow (BM) measured by MR spectroscopy
Interim efficacy: Bone mineral density as assessed by DEXA scan measured in grams per cubic centimeter with resulting Z score | From inclusion to 12 months of study treatment
  Change in bone mineral density (BMD) measured by DEXA scan measured in grams per cubic centimeter with resulting Z score.
Interim efficacy: Body composition as assessed by DEXA scan presented as whole body bone mass and soft tissue composition | From inclusion to 12 months of study treatment
  Change in body composition measured by DEXA scan presented as whole body bone mass and soft tissue composition with ratios of lean mass, body fat, and bone mass.
Interim efficacy: Gut microbiota composition as assessed by 16S rRNA sequencing | From inclusion to 4 months of study treatment
  Change in gut microbiota by 16S rRNA sequencing or whole genome sequencing of intestinal bacteria.
Interim efficacy: Gut microbiota composition as assessed by 16S rRNA sequencing | From inclusion to 12 months of study treatment
  Change in gut microbiota by 16S rRNA sequencing or whole genome sequencing of intestinal bacteria.
Interim efficacy: Small intestinal permeability as assessed by urine-lactulose/mannitol measurement and ion chromatography | From inclusion to 4 months of study treatment
  Change in small intestinal permeability by functional assessment by urine-lactulose/mannitol measurement and ion chromatography or by indirect assessment by qPCR and 16S rRNA sequencing of whole blood.
Interim efficacy: Epigenetic regulation as assessed by levels of 5-mC and 5-hmC | From inclusion to 4 months of study treatment
  Change in DNA methylation and hydroxymethylation (5-mC and 5-hmC) patterns in hematopoietic cells by global 5-hmC/5-mC assessment and EPIC arrays.
Interim efficacy: Epigenetic regulation as assessed by levels of 5-mC and 5-hmC | From inclusion to 12 months of study treatment
  Change in DNA methylation and hydroxymethylation (5-mC and 5-hmC) patterns in hematopoietic cells by global 5-hmC/5-mC assessment and EPIC arrays.
Interim efficacy: Gene expression as assessed by RNA sequencing | From inclusion to 4 months of study treatment
  Change in RNA expression in hematopoietic cells and BM adipocytes.
Interim efficacy: Gene expression as assessed by RNA sequencing | From inclusion to 12 months of study treatment
  Change in RNA expression in hematopoietic cells and BM adipocytes.
Interim efficacy: Protein profiles as assessed by proteomics | From inclusion to 4 months of study treatment
  Change in protein profiles in hematopoietic cells and BM adipocytes by proteomics.
Interim efficacy: Protein profiles as assessed by proteomics | From inclusion to 12 months of study treatment
  Change in protein profiles in hematopoietic cells and BM adipocytes by proteomics.
Interim efficacy: Response and disease progression as according to the IWG response criteria in myelodysplastic neoplasms | From inclusion to 12 months of study treatment
  Rates of response and disease progression as according to the International Working Group (IWG) response criteria in myelodysplastic neoplasms.
Interim efficacy: Bone marrow niche factor levels as assessed by ELISA | From inclusion to 4 months of study treatment
  Change in niche factors in bone marrow by ELISA.
Interim efficacy: Bone marrow niche factor levels as assessed by ELISA | From inclusion to 12 months of study treatment
  Change in niche factors in bone marrow by ELISA.
Interim efficacy: Cytokine levels as assessed by ELISA | From inclusion to 4 months of study treatment
  Change in cytokine levels in peripheral blood and bone marrow plasma by ELISA.
Interim efficacy: Cytokine levels as assessed by ELISA | From inclusion to 12 months of study treatment
  Change in cytokine levels in peripheral blood and bone marrow plasma by ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Grønbæk, Professor, MD, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Copenhagen N, Denmark